CLINICAL TRIAL: NCT00748722
Title: Pre-Operative Imaging of Abdominal Wall Perforators Using CT Angiography for DIEP Breast Reconstruction
Brief Title: Pre-Operative Imaging of Abdominal Wall Perforators Using CT Angiography
Acronym: DIEP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Yoav Barnea, MD, Tel Aviv Medical Center
Other Study IDs: TASMC-08-YB-0181-CTIL
Record Dates: First submitted 2008-07-15; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Breast Reconstruction
Keywords: Breast reconstruction; Perforator flaps; CT Angiography
MeSH Terms: interventions — Computed Tomography Angiography; Thyroid Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Female patients, age 18-60 years, suitable for breast reconstruction using the lower abdominal tissue.
  Interventions: Device: CT Angiography

INTERVENTIONS:
Device: CT Angiography — Injection of contrast material (iodine)
  Other Names: Iodine

SUMMARY:
Abdominal donor-site flaps, including the transverse rectus abdominis musculocutaneous (TRAM) and deep inferior epigastric artery perforator flaps(DIEP), are standard in autologous breast reconstruction. With significant variation in the vascular anatomy of the abdominal wall, preoperative imaging is essential for preoperative planning and reducing intraoperative error.

The quest continues for optimal preoperative assessment. Computed tomographic angiography has recently been proposed as a noninvasive modality for this purpose. It provides the location of the perforator vessels, diameter and anatomic course in regards to the rectus muscle.

In this study we will perform preoperative lower abdominal computed tomographic angiography in DIEP flap breast reconstruction patients.

DETAILED DESCRIPTION:
Abdominal donor-site flaps, including the transverse rectus abdominis musculocutaneous (TRAM) and deep inferior epigastric artery perforator flaps(DIEP), are standard in autologous breast reconstruction. With significant variation in the vascular anatomy of the abdominal wall, preoperative imaging is essential for preoperative planning and reducing intraoperative error.

The quest continues for optimal preoperative assessment. Computed tomographic angiography has recently been proposed as a noninvasive modality for this purpose. It provides the location of the perforator vessels, diameter and anatomic course in regards to the rectus muscle.

In this study we will perform preoperative lower abdominal computed tomographic angiography in DIEP flap breast reconstruction patients.

We plan to study 20 patients, eligible for lower abdominal-based breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-60 years
* Appropriate for lower abdominal based breast reconstruction.
* Consented the use of CT Angiography

Exclusion Criteria:

* Age under 18 years or over 60.
* Pregnant women
* Allergy to iodine

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients, age 18-60 years eligible for lower abdominal breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
1 year from starting date | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Barnea, MD, Study Chair — Tel Aviv Medical Center; Arie Blachar, MD, Principal Investigator — Tel Aviv Medical Center; Eyal Gur, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel-Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Rozen WM, Palmer KP, Suami H, Pan WR, Ashton MW, Corlett RJ, Taylor GI. The DIEA branching pattern and its relationship to perforators: the importance of preoperative computed tomographic angiography for DIEA perforator flaps. Plast Reconstr Surg. 2008 Feb;121(2):367-373. doi: 10.1097/01.prs.0000298313.28983.f4. PMID 18300951
- [Result] Rozen WM, Phillips TJ, Ashton MW, Stella DL, Gibson RN, Taylor GI. Preoperative imaging for DIEA perforator flaps: a comparative study of computed tomographic angiography and doppler ultrasound. Plast Reconstr Surg. 2008 Jan;121(1 Suppl):1-8. PMID 18213740